CLINICAL TRIAL: NCT02708589
Title: The Effects of Probiotic Supplementation on Anthropocentric, Nutrients Status, Inflammation, GI Hormones, Quality of Life, and Microflora in Patients Undergoing Gastric Bypass Surgery
Brief Title: The Effects of Probiotic Supplementation on the Results of Gastric Bypass Surgery
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Associate Prof, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 600
Record Dates: First submitted 2016-03-01; First posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Gastric Bypass Surgery
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- probiotic (Active Comparator): the probiotics capsules contain 7 strains of friendly bacteria (Lactobacillus casei, Lactobacillus rhamnosus, Streptococcus thermophilus, Bifidobacterium breve, Lactobacillus acidophilus, Bifidobacterium longum, and Lactobacillus bulgaricus) and prebiotic (fructooligosaccharide).
  Interventions: Dietary Supplement: probiotic
- Placebo (Placebo Comparator): Placebo capsules have identical appearance to probiotic capsules and contain Maltodextrin.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: probiotic
  Arms: probiotic
Other: Placebo
  Arms: Placebo

SUMMARY:
In this study, patients undergoing the bariatric surgery will be assigned to take either probiotic capsules or placebos from 1 month before surgery to 3 months after the surgery. Their anthropometric and biochemical measurements will be assessed every 3-6 months, and will be compared in two groups.

ELIGIBILITY:
Inclusion Criteria:

* BMI> 40 or >35 plus other morbidities
* Undergoing the gastric bypass surgery
* Willing to participate in the study

Exclusion Criteria:

* History of any chronic GI or kidney disorders, malignancies, or immune deficiencies
* Taking any immunomodulatory or immunosuppressor medications
* Taking Antibiotics from 4 weeks before and during the intervention
* Being on special diet such as vegetarian diet
* Doing as a professional Athlete
* Pregnancy and Lactation

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
weigh of the participants will be measured in Kg. | 3 months after surgery

SECONDARY OUTCOMES:
serum level of vitamin B12 (mg/dl) | 3 months after surgery
serum level of vitamin B12 (mg/dl) | 12 months after surgery
serum level of vitamin D(ng/ml) | 3 months after surgery
serum level of vitamin D (ng/ml) | 12 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- NNFTRI clinic, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Mokhtari Z, Karbaschian Z, Pazouki A, Kabir A, Hedayati M, Mirmiran P, Hekmatdoost A. The Effects of Probiotic Supplements on Blood Markers of Endotoxin and Lipid Peroxidation in Patients Undergoing Gastric Bypass Surgery; a Randomized, Double-Blind, Placebo-Controlled, Clinical Trial with 13 Months Follow-Up. Obes Surg. 2019 Apr;29(4):1248-1258. doi: 10.1007/s11695-018-03667-6. PMID 30612325
- [Derived] Karbaschian Z, Mokhtari Z, Pazouki A, Kabir A, Hedayati M, Moghadam SS, Mirmiran P, Hekmatdoost A. Probiotic Supplementation in Morbid Obese Patients Undergoing One Anastomosis Gastric Bypass-Mini Gastric Bypass (OAGB-MGB) Surgery: a Randomized, Double-Blind, Placebo-Controlled, Clinical Trial. Obes Surg. 2018 Sep;28(9):2874-2885. doi: 10.1007/s11695-018-3280-2. PMID 29725975